CLINICAL TRIAL: NCT03531346
Title: A 12-month Prospective Study of Tear Osmolarity in Contact Lens Wearers Refitted With Daily Disposable Soft Contact Lenses
Brief Title: Tear Osmolarity Changes in Habitual Contact Lens Wearers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Collaborators: Wrocław University of Science and Technology (Other)
Responsible Party: Principal Investigator, Izabela Garaszczuk, Principal Investigator, Researcher, Optometrist, University of Valencia
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 642760
Record Dates: First submitted 2018-05-08; First posted 2018-05-21 (Actual); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Tear Film Hyperosmolarity
Keywords: Tear film; Tear osmolarity; Contact lenses

STUDY DESIGN:
Who Masked: Participant
Masking Description: Subjects were masked with respect to the lens type.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyperosmolarity group (Experimental): Healthy, young, habitual contact lens wearers with initial increased tear osmolarity (hyperosmolarity)
  Interventions: Other: Daily-disposable soft contact lens
- Normal osmolarity (Experimental): Healthy, young, habitual contact lens wearers with initial tear osmolarity reported as normal
  Interventions: Other: Daily-disposable soft contact lens

INTERVENTIONS:
Other: Daily-disposable soft contact lens — Subjects were refitted with Silicone-Hydrogel (Delefilcon A) or Hydrogel (Omafilcon A) daily-disposable soft contact lenses based on their fit, reported comfort and tear film surface quality.

SUMMARY:
Tear osmolarity refers to the amount of osmotically active particles in tears and has been reported as one of the best diagnostic test for dry eye disease. Our research focused on following changes in tear osmolarity and ocular symptoms in the time-course of one year after refitting habitual contact lens wearers or fitting novices with modern daily disposable soft contact lenses. Fifty-six contact lens wearers aged (mean ± standards deviation) 26 ± 4 y/o were refitted with Silicone-Hydrogel (Delefilcon A) or Hydrogel (Omafilcon A) lenses.

Study included seven visits: baseline measurement before the study, two visits for contact lens fit and control and follow-up measurements after three, six, and 12 months of contact lens wear followed by measurements on bare eye according to the baseline scheme (post-study visit).

An impedance-based osmometer was used to collect samples from the lower tear meniscus. A standard Ocular Surface Disease Index (OSDI) questionnaire was used to monitor subject-reported ocular symptoms. Statistically significant differences were noted in tear osmolarity in the time course of the study for both eyes.

An improvement in tear osmolarity was most prevalent among subjects with high initial tear osmolarity. Low osmolarity levels were maintained after the study.

The findings of this prospective study will reveal that habitual contact lens wearers or novices may benefit from refitting with modern daily disposable soft contact lenses.

DETAILED DESCRIPTION:
Tear osmolarity refers to the amount of osmotically active particles in tears and is defined as the number of osmoles per litre of solution. It is mostly determined by the electrolytes of the aqueous component of tears and less significantly by proteins and sugars. It has been described as a single clinical measure that gives insight into the balance between tear production, evaporation, drainage and absorption of tears. Studies support the use of tear osmolarity as the best single diagnostic test for dry eye disease (DED) and the objective numerical measure for diagnosing, grading severity, and managing DED. Clinical application was facilitated after introducing a chip-based osmometer (TearLab® Osmolarity System, TearLab Corp, San Diego, California, USA)7, which allows collection of a relatively small sample of 50 nL from the inferior tear meniscus and automatic determination of tear osmolarity, based on the sample's conductivity.

The osmolarity of 308 mOsm/L is considered to be the most sensitive threshold to distinguish normal from mild/moderate forms of DED and 315 mOsm/L the most specific cut off. Also the inter-eye difference in osmolarity increases with DED severity and beyond the threshold of 8 mOsm/L it is considered an indication of the loss of tear film homeostasis. In normal subjects this variation between eyes is around 6.9 ± 5.9 mOsm/L. Tear film with a contact lens undergoes biophysical and biochemical changes, which have the potential to influence tear function and impact comfort and contact lens tolerance. Many factors have been associated with lowering of comfort and changes in tear dynamics during lens wear, however the literature is divided over whether or not contact lens wear increases, or has no effect on tear osmolarity.

The differences in reported values are likely a function of the wearer's ability to maintain tear film homeostasis, overcoming the drying effect of contact lenses.

Tear osmolarity was reported as the least variable of all the common signs across a clinically relevant timeframe, and was the only sign to reduce its variation upon application of effective therapy.

Tear hyperosmolarity is a clinical starting point in the pathogenesis of DED, responsible for ocular surface damage, both directly and by initiating a chain of inflammatory responses leading to ocular surface damage. Contact lens wear increases the risk of developing DED from between 2.01 and 2.96 times. Wearers are much more likely to report discomfort, mostly described as dryness and end of day dryness, than non-wearers and this factor remains the single largest cause of contact lens wear discontinuation. However, a multifactorial nature of DED, disguised as a lack of association between clinical signs and reported symptoms, leads to underlying cause of contact lens discomfort and remains poorly understood. Contact lens related DED may be explained by increased tear film thinning times resulting in increased tear film osmolality or by the loss of corneal sensation particularly associated with long-standing wear of hard and extended-wear contact lenses. Lowered corneal sensitivity leads to decreased tear secretion in response to reflex stimuli presumably causing an increase in tear osmolarity. Tear hyperosmolarity has been reported in daily and extended wear of both soft and hard contact lens wearers, especially in symptomatic subjects. Extended-wear soft contact lenses can decrease corneal sensitivity more than daily-wear soft contact lenses. A significant increase in tear osmolarity could not be confirmed in subjects wearing daily disposable soft contact lenses.

Few studies have been conveyed to investigate the longitudinal effects of soft contact lens wear on ocular physiology. These studies generally focused on different lens designs and oxygen permeability and their impact on the ocular surface morphology, tear stability or ocular surface sensory function.

Changes in ocular physiology during contact lens wear are evident, however the effect of modern daily disposable contact lens on tear film osmolarity still remains unknown. In the last decade significant advancements have been made in both contact lens technology and DED diagnosis. Therefore, further evaluation of the influence of modern contact lenses on ocular physiology is necessary.

The hypothesis of this research is that the wear of modern daily disposable soft contact lenses maintains tear film osmolarity in compliant habitual contact lens wearers or novices. Hence, the objective was to investigate the potential changes in tear osmolarity experienced during the wear of such lenses across a period of 12 months.

The study adhered to the tenets of the Declaration of Helsinki. Informed consent was obtained from each participant after the nature and possible consequences of the study were explained. The study recruited 60 healthy young novices or habitual contact lens wearers (41 F and 19 M), aged (mean ± standard deviation) 26 ± 4 y/o, ranging from 20 to 37 y/o. Habitual contact lens users were advised to cease wearing their lenses and instilling ophthalmic solutions at least three days prior to commencing the study.

This was to ensure subjects previously wearing different types of contact lenses achieved a more consistent baseline (bare eye) result. Subjects were also requested to present an up-to-date optical prescription. Exclusion criteria were signs and symptoms of severe eye dryness, inflammation or substantial tear flow impairment and any systemic disorders known to compromise the ocular surface or tear film quality. Additionally, subjects were excluded if demonstrated at least two out of the following signs of DED: OSDI higher than 23, conjunctival staining higher or equal to 2 or/and corneal staining higher or equal to 2 present (Efron grading scale) and fluorescein tear film break-up time of less than 7 seconds. The refractive error was limited to ±5.00 spherical and ±0.75 cylindrical diopters, as the spherical equivalent of the correction was provided

The study protocol consisted of a qualifying visit (Baseline), contact lens fitting visit (following day - Day 2 visit), a control visit at 2 weeks and follow-up visits at 3 months, 6 months and 12 months post-refitting, followed by the visit for the post-study assessment after three days (post-study visit). Laboratory temperature (°C) and humidity (%Rh) were monitored with the thermo-hygrometry device (C3121, Comet, Czech Republic). Subjects could have an environmental adjusting period if they arrived at the laboratory directly from the outdoors. At each of the visits (except Day 2) OSDI questionnaire was filled-in by the participants to assess ocular symptoms during the last week preceding each visit and to distinguish symptomatic subjects.

Subjects with OSDI ≥ 13 were reported as symptomatic, as this is the reported threshold between healthy and mild/moderate DED subjects. The questionnaire was adapted to the subjects' native language. During the Baseline visit, together with OSDI, the review of medical history was performed including general and ocular health, refractive correction type, modality and refractive power, visual acuity (distance and near), the date of last eye examination and last medical examination, history of previous contact lens wear, family ocular history, allergies, medication, occupation, driving, visual display unit use, smoking and hobbies. This was followed by tear osmolarity measurements with TearLab Osmolarity System (TearLab Corp. San Diego, CA. Measurements performed at Baseline were used for qualifying subjects to the study and formed the baseline database for comparative analyses with the measurements performed at follow-up visits. Measurements at Baseline and post-study visit were performed at the same time of the day.

At Day 2 (the following day) subjects were fitted with Silicone-Hydrogel (Si-Hy, Delefilcon A) or Hydrogel (Hy, Omafilcon A) daily disposable soft contact lenses.

Newly-fitted lens was chosen based on contact lens fit, reported subjective comfort after 4 hours of wear and pre-lens tear film surface quality. Contact lens fit assessment included contact lens centration, corneal coverage, horizontal lag, blink movement, push-up test and the binocular corrected visual acuity rating for distance and near vision.

A supply of contact lenses was provided for each subject, with the instruction to wear the lenses for any five days per week, minimum eight hours and up to 12 hours per day. The same wearing schedule was followed for the whole duration of the study.

All subjects were fully instructed on insertion, safe removal and lens care together with the given written instructions. The purpose of the 2-week control visit was to ensure good contact lens performance, comfort and fit and to qualify subjects for 12 months of contact lens wear. At three-, six- and 12-month visits subjects were advised to wear their contact lenses at least five hours prior to attending. The protocol for these follow-up visits included OSDI questionnaire filled in during an environmental adjusting break, osmolarity measurements on bare eye and ocular anterior surface check-up with the slit-lamp biomicroscope to assess ocular surface health.

Tear osmolarity was measured for both eyes of each subject from the inferior lateral tear meniscus. Electronic check cards calibration of the instrument was performed daily according to the manufacturer's instruction. The calibration using a control solution was performed every time a new box of test cards was opened.

The device was powered for the whole duration of the study where diagnostic pens were kept fully charged. The device and the test cards were stored in the laboratory in which the measurements were conducted. The same diagnostic pen was used for all measurements, starting the assessment, every time, with the right eye. Samples were collected by the same experienced researcher from the eye without contact lens, 10 minutes after subject taking the lenses off. Subjects were asked to sit with their chin tilted slightly upward and eyes directed toward the ceiling. The tip of the pen was positioned just above the lower eyelid and gently applied to the thin line of tears on the lower eyelid margin. Care was taken not to induce reflex lacrimation. After successful collection, the values were recorded. At least two measurements for each eye were performed. If the results were not consistent (differed more than 10 mOsm/L), the third measurements was conducted. The tear film osmolarity was measured at the Baseline, three-month, six-month, 12-months and the post-study visits.

ELIGIBILITY:
Inclusion Criteria:

* The refractive error limited to ±5.00 spherical and ±0.75 cylindrical diopters
* Subjects with up-to-date optical prescription

Exclusion Criteria:

* Signs and symptoms of severe eye dryness or inflammation
* Substantial tear flow impairment
* Any systemic or ocular disorder known to compromise the ocular surface or tear film quality.
* At least two out of the following signs of dry eye disease:

  * Ocular Surface Disease Index higher or equal to 23,
  * Conjunctival staining higher or equal to 2 or/and corneal staining higher or equal to 2 (graded with Efron grading scale)
  * Fluorescein tear film break-up time shorter than 7 seconds.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-10-06 (Actual); Primary Completion 2016-12-16 (Actual); Study Completion 2017-12-07 (Actual)

PRIMARY OUTCOMES:
Tear film osmolarity | 3 months
  Tear film osmolarity measured after 3-months of wearing newly-fitted contact lenses

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garaszczuk IK, Mousavi M, Szczesna-Iskander DH, Cervino A, Iskander DR. A 12-month Prospective Study of Tear Osmolarity in Contact Lens Wearers Refitted with Daily Disposable Soft Contact Lenses. Optom Vis Sci. 2020 Mar;97(3):178-185. doi: 10.1097/OPX.0000000000001488. PMID 32168240